CLINICAL TRIAL: NCT06245798
Title: Liver Resection for Patients With Hepatocellular Carcinoma and Clinically Significant Portal Hypertension: A Chinese Multicentre Retrospective Cohort Study
Brief Title: Liver Resection for Patients With Hepatocellular Carcinoma and Clinically Significant Portal Hypertension
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Tangdu Hospital
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Hepatic Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- liver resection
- transarterial chemoembolisation
  Interventions: Procedure: transarterial chemoembolisation

INTERVENTIONS:
Procedure: transarterial chemoembolisation — During transarterial chemoembolisation（TACE）, a vascular catheter was selectively inserted into the tumour-feeding artery with an injection containing a mixture of doxorubicin (10-50 mg) and lipiodol (2-20 mL), followed by embolisation using gelatin sponge particles. TACE was repeated when residual viable tumours were confirmed or new lesions developed in patients with adequate liver function
  Groups: transarterial chemoembolisation

SUMMARY:
Clinically significant portal hypertension limits the therapeutic options for hepatocellular carcinoma (HCC), which is closely associated with patient prognosis. HCC patients with CPSH are heterogeneous and treatment allocation remains controversial. The aim of this study was to compare the survival benefits of liver resection (LR) and transarterial chemoembolisation (TACE) in these populations.

ELIGIBILITY:
Inclusion Criteria:

* HCC patients treated conventional liver resection or transarterial chemoembolisation

Exclusion Criteria:

* (1) presence of types III/IV portal vein tumour thrombosis (PVTT), hepatic artery, biliary duct or inferior vena cava invasion; (2) presence of extrahepatic spread (EHS); (3) underwent previous treatments; (4) Eastern Cooperative Oncology Group Performance Status (ECOG-PS) >1; (5) diffuse tumor nodules; (6) combined with other tumours or severe cardiac, cerebral, and renal insufficiency; (7) non-Clinically significant portal hypertension（CSPH）, and (8) absence of baseline information

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study data were extracted from a nationwide database of HCC patients treated at 15 Chinese centres between January 2012 and December 2022. We included patients who were diagnosed with HCC according to the American Association for the Study of the Liver Disease/European Association for the Study of the Liver Guidelines and who received conventional liver resection or transarterial chemoembolisation
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
overall survival rate | 5 year
  overall survival rate

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tangdu hospital, Xi'an, Shaanxi
  - Xijing hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No